CLINICAL TRIAL: NCT06294756
Title: Effects of Sulfurous Thermal Waters Inhalations on Long-COVID Syndrome: a Double-blinded, Interventional, Randomized Case-control, Pilot Study on a Spa Centered Rehab Program
Brief Title: Sulfureous Water Therapy in Viral Respiratory Diseases
Acronym: STWandRVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Università degli studi di Roma Foro Italico (Other); Queen Mary University of London (Other); Bios Prevention Srl (Unknown)
Responsible Party: Principal Investigator, Mario Fontana, Associate Professor of Biochemistry, Resident physician, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: acquealbuleroma1; AR1221816703484E (Other Grant/Funding Number: La Sapienza University, Rome, Italy)
Record Dates: First submitted 2024-02-09; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Long-COVID; Post COVID-19 Condition; Chronic COVID-19 Syndrome; Post Acute Sequelae of COVID-19
Keywords: LONG-COVID; spa; Inhalation therapy; Sulfurous thermal water; H2S; Nasal microbiome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: The study is a double-blind, interventional, randomized case-control, pilot trial assessing the efficacy of sulfureous thermal water (STW) inhalations in patients diagnosed with long-COVID. The eligible subjects were randomized in a 1:1 ratio to either: active (STW) or placebo (SDW) group for the inhalation therapy and tested at 3 timepoints: Visit 1 (prior treatment), Visit 2 (just after treatment) , Visit 3 (3 months after treatment).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither the participants nor any of the medical researchers or laboratory staff involved in the screening, enrolment, clinical evaluation, monitoring, and laboratory as well as statistics of the participant's analyses were aware of the study intervention received (STW vs SDW). A randomization list (1:1 active vs placebo) was created prior to recruiting. The inhalation assistant randomized the participant according to the list and administered the intervention. Therefore, the inhalation assistant was unblinded to the treatment assigned but blinded to the medical condition of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long covid patients undergoing inhalations with sulfurous thermal water (STW) (Active Comparator): Adult Outpatients aged 18-75, presenting to the spa facility with an independent prescription of inhalation therapy with sulfurous water for post-COVID respiratory issues.
  Active arm treatment consisted of 12 consecutive sessions of sulfurous thermal water (STW) from Visit 1 for 12 days.
  Re-assessment of study analyses was performed on Visit 2 after, 14 days from Visit 1. The follow-up (Visit 3) was 90 days after Visit 1.
  Interventions: Other: Inhalation of Sulfurous Thermal Water
- Long covid patients undergoing inhalations with Sterile Distilled non-pyrogenic Water (SDW) (Placebo Comparator): Adult Outpatients aged 18-75, presenting to the spa facility with an independent prescription of inhalation therapy with sulfurous water for post-COVID respiratory issues. Placebo arm treatment consisted of 12 consecutive sessions of Sterile Distilled non-pyrogenic Water (SDW) from Visit 1 for 12 days.
  Re-assessment of study analyses was performed on Visit 2 after, 14 days from Visit 1. The follow-up (Visit 3) was 90 days after Visit 1.
  Interventions: Other: Inhalation of Sterile Distilled non-pyrogenic Water

INTERVENTIONS:
Other: Inhalation of Sulfurous Thermal Water — Active Inhalation protocol based on 12 consecutive sessions, 20 minutes each, once a day from Visit 1 through a conventional thermal water aerosolization Faset™system (Faset Spa, Trezzano sul Naviglio, Milan, Italy) delivering particles of TW with a diameter between 0.6 µm <MMAD < 5 µm. Treatment consisted of 10 minutes of warm steam and 10 minutes of aerosol inhalation with nasal prongs.
  Other Names: STW aerosol; STW steam inhalation
  Arms: Long covid patients undergoing inhalations with sulfurous thermal water (STW)
Other: Inhalation of Sterile Distilled non-pyrogenic Water — Placebo Inhalation protocol based on 12 consecutive sessions, 20 minutes each, once a day from Visit 1 through a modified thermal water aerosolization Faset™system, previously disconnected from the hydraulic circuit that supplied TW and connected to non-pyrogenic sterile water reservoirs (Highly depurated water- Pharmaceutical grade FU-for external and internal use, Makeitlab, Canosa di Puglia, BT, Italy). Treatment consisted of 10 minutes of warm steam and 10 minutes of aerosol inhalation with nasal prongs delivering particles of SDW with a diameter between 0.6 µm <MMAD < 5 µm.
  Other Names: SDW aerosol; SDW steam inhalation
  Arms: Long covid patients undergoing inhalations with Sterile Distilled non-pyrogenic Water (SDW)

SUMMARY:
The goal of this double-blind, interventional, randomized case-control, pilot trial is to evaluate the effects of active sulfurous (STW) versus placebo (SDW) inhalations on blood test parameters, serum inflammatory cytokines, spirometry data, as well as qualitative and quantitative changes in the nasal microbiome of subjects affected by long Covid.

The main questions it aims to answer are:

* if STW inhalations are effective on respiratory issues due to long covid compared to the placebo inhalation (SDW)
* if STW inhalations are effective on long covid related fatigue issues compared to the placebo inhalation (SDW)
* if H2S inhaled with STW is effective in modulating (decreasing) cytokines which are related to long covid cytokine storm compared to placebo inhalation with no H2S (SDW)
* if STW inhalation modify nasal microbiome both from a qualitative and quantitative point of view respect to placebo inhalation (SDW) Participants will be randomly assigned to active inhalations (STW) or placebo inhalations (SDW) arm and subjected to 12 consecutive sessions of 20 minutes.

Both arms will be tested for:

* cytokines and inflammatory markers concentration (IL1b, IL6, ACE, GSS, S100B, Hs-CRP)
* spirometry (resting, forced, DLCO)
* exertion response (6 minutes walking test)
* nasal microbiome sampling at visit 1 (enrolment), at visit 2(right after the inhalation treatment) and at visit 3 (3 months after treatment).

Researchers will compare results reported by STW to those of SDW group to see if significative differences are detectable.

DETAILED DESCRIPTION:
The study is a double-blind, interventional, randomized case-control, pilot trial assessing the efficacy of sulfureous thermal water (STW) inhalations in patients diagnosed with long-COVID. The study was performed from May to October 2023 at the Acque Albule spa facility, Terme di Roma, Tivoli Terme, Rome, Italy. The SPA-center rehab program included 12 consecutive sessions for 20 minutes each from day 1 for 12 days. Re-assessment of study analyses was performed on day 14 after (Visit 2). The follow-up (Visit 3) was 90 days after Visit 1.

Eligible subjects were adult outpatients, presenting to the spa facility with an independent prescription of inhalation therapy with sulfurous water for post-COVID respiratory issues. The participants had previously tested positive in certified PCR screening for SARS-Cov-2 infection (data from the Regional Archive of Health Service for SARS-Cov-2 Infection) and, at the time of the study, had a positive diagnosis of long-COVID syndrome with pulmonary involvement.

Neither the participants nor any of the medical researchers or laboratory staff involved in the screening, enrolment, clinical evaluation, monitoring, and laboratory as well as statistics of the participant's analyses were aware of the study intervention received (STW vs SDW). A randomization list (1:1 active vs placebo) was created prior to recruiting. The inhalation assistant randomized the participant according to the list and administered the intervention. Therefore, the inhalation assistant was unblinded to the treatment assigned but blinded to the medical condition of the participants.

At each session of treatment delivered at Visit 1 and Visit 2, participants were tested for SARS-Cov-2 infection, underwent resting plus forced spirometry and alveolar-capillary diffusion of carbon monoxide (DLCO) spirometry, and performed the the six minutes walking test (6MWT). St George Respiratory Questionnaire (SGQ) used to determine the impact of pulmonary impairment on the quality of life was completed at Visit 1 and Visit 3, patient satisfaction survey was submitted to participants at Visit 3 only. Moreover, blood samples for routine analysis, urine sample collections, and nasal swabs for microbiome sampling were collected at each visit. At the end of Visit 1 (screening/enrolment day), the eligible subjects were randomized in a 1:1 ratio to either: active (STW) or placebo (SDW) group for the inhalation therapy. Both active and controls underwent inhalation therapy once a day for 12 days (from day 1).

ELIGIBILITY:
Inclusion Criteria:

* · Adults aged from 18 to 75.

  * Willing and capable of giving informed consent.
  * Participants with smoking habits or not
  * Participants with COVID vaccination or not
  * Negative to Sars-Cov2 rapid swabs at screening visit
  * Certified previous Sars Cov2 infection (Regional Public Health Service archives of Sars Cov2 infection)
  * Certified diagnosis of long COVID (post-infective onset symptoms only, lasting more than 4 months since swab negativisation).
  * Any severity of Covid symptoms during acute infection (Home care, ICU admission, ventilation)
  * Participants treated with inhaled bronchodilators or not.
  * Willing and able to comply with scheduled visits, laboratory tests, and other study procedures.

Exclusion Criteria:

* · Obesity (BMI>32).

  * Walking impairment.
  * Pre-existing other comorbidities affecting the airways (e.g., asthma, rhinitis, etc.).
  * Therapy with inhaled, IV, or IM steroids.
  * Pre-existing diagnosis of depression, psychological or psychiatric disorders.
  * Patients currently recruited to other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
To determine whether Sulfurous Thermal water (STW) inhalations may have effects on post covid-pulmonary sequelae assessing changes in pulmonar functionality through spirometric parameters. | Day1
  To assess the prior treatment whole pulmonary functionality by spirometry and DLCO spirometry
To determine whether Sulfurous Thermal water (STW) inhalations may have effects on post covid-pulmonary sequelae assessing changes in pulmonar functionality through spirometric parameters. | Day 14
  To assess the whole pulmonary functionality at 14 days since inhalations start by spirometry and DLCO spirometry
To determine whether Sulfurous Thermal water (STW) inhalations may have effects on post covid-pulmonary sequelae assessing changes in pulmonar functionality through spirometric parameters | Day 90
  To assess the whole pulmonary functionality at 90 days since inhalations start by spirometry and DLCO spirometry.
To determine whether Sulfurous Thermal water (STW) inhalations can improve the cardiopulmonary response to physical exertion measured as SpO2, Heart rate, Borg score and traversed meters in patients affected by long COVID | Day 1
  To assess the cardiopulmonary response to physical exertion prior inhalations therapy with the six minutes walking test (6MWT)
To determine whether Sulfurous Thermal water (STW) inhalations can improve the cardiopulmonary response to physical exertion measured as SpO2, Heart rate, Borg score and traversed meters in patients affected by long COVID | Day 14
  To assess the cardiopulmonary response involved during physical exertion at 14 days since inhalations start with the six minutes walking test (6MWT)
To determine whether Sulfurous Thermal water (STW) inhalations can improve the cardiopulmonary response to physical exertion measured as SpO2, Heart rate, Borg score and traversed meters in patients affected by long COVID | Day 90
  To assess the cardiopulmonary response to physical exertion at 90 days since inhalations start with the six minutes walking test (6MWT)

SECONDARY OUTCOMES:
To assess if H2S present in STW can interfere with concentration of inflammatory markers ( as IL1B, IL-6, ACE, S100B, GSS, Hs-CRP) typically alterated in long covid patients. | Day 1
  To assess serum inflammatory responses prior inhalations treatment by determining IL-6, IL-1β, S100B, GSS, ACE serum concentration
To assess if H2S present in STW can interfere with concentration of inflammatory markers ( as IL1B, IL-6, ACE, S100B, GSS, Hs-CRP) typically alterated in long covid patients. | Day 14
  To assess serum inflammatory responses at 14 days since inhalations treatment start by determining IL-6, IL-1β, S100B, GSS, ACE serum concentration
To assess if H2S present in STW can interfere with concentration of inflammatory markers ( as IL1B, IL-6, ACE, S100B, GSS, Hs-CRP) typically alterated in long covid patients. | Day 90
  To assess serum inflammatory responses at 90 days since inhalations treatment start by determining IL-6, IL-1β, S100B, GSS, ACE serum concentration
to assess whether thermal water inhalation with sulfurous water may determine qualitative and quantitative changes of the nasal microbiome by assessing alpha and beta diversity after nasal sample collection | Day 1
  Collection with swabs and 16SrDNA analysis of the nasopharyngeal secretions prior inhalations treatment.
to assess whether thermal water inhalation with sulfurous water may determine qualitative and quantitative changes of the nasal microbiome by assessing alpha and beta diversity after nasal sample collection | Day 14
  Collection with swabs and 16S rDNA analysis of the nasopharyngeal secretions at 14 days since inhalations treatment start
to assess whether thermal water inhalation with sulfurous water may determine qualitative and quantitative changes of the nasal microbiome by assessing alpha and beta diversity after nasal sample collection | Day 90
  Collection with swabs and 16S rDNA analysis of the nasopharyngeal secretions at 90 days since inhalations treatment start

OTHER OUTCOMES:
to assess whether thermal water inhalation determine changes in the perceived impact of respiratory related impairment on the quality of life (Qol) through a validate Saint George respiratory questionnaire | Day 1
  Impact of post covid respiratory-related impairment on the quality of life prior treatment is evaluated using the Saint George respiratory questionnaire (SGRQ)
to assess whether thermal water inhalation determine changes in the perceived impact of respiratory related impairment on the quality of life (Qol) through a validate Saint George respiratory questionnaire | Day 90
  90 days after treatment Impact of post covid respiratory-related impairment on the quality of life is evaluated using the Saint George respiratory questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Fontana, Prof, MD, Study Chair — La Sapienza, University of Rome; Serena Crucianelli, MD, Principal Investigator — La Sapienza, University of Rome; Alessia Mariano, PhD, Principal Investigator — La Sapienza, University of Rome
Locations (1):
- Acque Albule, Terme di Roma, Tivoli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fowora MA, Aiyedogbon A, Omolopo I, Tajudeen AO, Olanlege A-L, Abioye A, Akintunde GB, Salako BL. Effect of nasal carriage of Bacillus species on COVID-19 severity: a cross-sectional study. Microbiol Spectr. 2024 Feb 6;12(2):e0184323. doi: 10.1128/spectrum.01843-23. Epub 2024 Jan 9. PMID 38193730
- [Result] Davis HE, McCorkell L, Vogel JM, Topol EJ. Long COVID: major findings, mechanisms and recommendations. Nat Rev Microbiol. 2023 Mar;21(3):133-146. doi: 10.1038/s41579-022-00846-2. Epub 2023 Jan 13. PMID 36639608
- [Result] Huerne K, Filion KB, Grad R, Ernst P, Gershon AS, Eisenberg MJ. Epidemiological and clinical perspectives of long COVID syndrome. Am J Med Open. 2023 Jun;9:100033. doi: 10.1016/j.ajmo.2023.100033. Epub 2023 Jan 18. PMID 36685609
- [Result] Low RN, Low RJ, Akrami A. A review of cytokine-based pathophysiology of Long COVID symptoms. Front Med (Lausanne). 2023 Mar 31;10:1011936. doi: 10.3389/fmed.2023.1011936. eCollection 2023. PMID 37064029
- [Result] Ribeiro Carvalho CR, Lamas CA, Chate RC, Salge JM, Sawamura MVY, de Albuquerque ALP, Toufen Junior C, Lima DM, Garcia ML, Scudeller PG, Nomura CH, Gutierrez MA, Baldi BG; HCFMUSP Covid-19 Study Group. Long-term respiratory follow-up of ICU hospitalized COVID-19 patients: Prospective cohort study. PLoS One. 2023 Jan 20;18(1):e0280567. doi: 10.1371/journal.pone.0280567. eCollection 2023. PMID 36662879
- [Result] Maccarone MC, Masiero S. Spa therapy interventions for post respiratory rehabilitation in COVID-19 subjects: does the review of recent evidence suggest a role? Environ Sci Pollut Res Int. 2021 Sep;28(33):46063-46066. doi: 10.1007/s11356-021-15443-8. Epub 2021 Jul 17. PMID 34273080
- [Result] Bazhanov N, Escaffre O, Freiberg AN, Garofalo RP, Casola A. Broad-Range Antiviral Activity of Hydrogen Sulfide Against Highly Pathogenic RNA Viruses. Sci Rep. 2017 Jan 20;7:41029. doi: 10.1038/srep41029. PMID 28106111
- [Result] Antonelli M, Donelli D. Respiratory rehabilitation for post-COVID19 patients in spa centers: first steps from theory to practice. Int J Biometeorol. 2020 Oct;64(10):1811-1813. doi: 10.1007/s00484-020-01962-5. Epub 2020 Jul 24. PMID 32710297
- [Result] Merenstein C, Bushman FD, Collman RG. Alterations in the respiratory tract microbiome in COVID-19: current observations and potential significance. Microbiome. 2022 Oct 5;10(1):165. doi: 10.1186/s40168-022-01342-8. PMID 36195943
- See also: Chemical composition of STW: Acque Albule, Terme di Roma — https://www.termediroma.org/pdf/analisi-chimico-fisico-2018.pdf